CLINICAL TRIAL: NCT04788589
Title: Effectiveness of Sedation and Ventilator Weaning Protocol - a Randomized Controlled Trial
Brief Title: Sedation and Ventilator Weaning Protocol in PICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Antonius Hocky Pudjiadi, SpA(K), Principal Investigator, Head of Pediatric Intensive Care Unit, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20030379
Record Dates: First submitted 2021-02-13; First posted 2021-03-09 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Mechanical Ventilation; Sedation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sedation and Ventilator Weaning Protocol (Experimental): Sedation: start midazolam 5-10 mins (max 3x). If MV 12 hrs-2d: Pain: morphine @2 hrs if needed (max 10mg/x). Sedation: midazolam @ 1-2 hrs if needed (max 10mg/x). If MV >2 d: morphine & midazolam drip (max 10mg/hr). MV weaning checklist @morning. Pass if no incr of sedation dose due to agitation, NMBAs, incr in ICP. Fail: reassessed tomorrow. Pain and SBS scores assessed @morning until extubation. Stop all sedation and analgetic for sedation. Continue analgetics for pain. Subjects monitored for 4 hrs. Assess pain and WAT-1 score. Pass (GCS of E3, tolerate sedation interruption for > 4 hrs): MV weaning protocol. Fail (Persistent anxiety/agitation, incr pain score, incr RR > 5 mins, SpO2 <88% >5 mins, acute heart dysrhythmia, >=2 signs of ARDS): sedation resumed ½ dose, up titrated.
  MV weaning: CPAP 5/PS < 7. Pass: No failure criteria for 2 hrs. Fail (Incr RR > 5 mins, SpO2 <88% > 5 mins, acute decr in GCS/acute heart dysrhythmia, >=2 signs of ARDS): previous MV setting.
  Interventions: Other: Sedation and ventilator weaning protocol
- Control (No Intervention): 1. Informed consent
  2. Randomization into groups
  3. Sedation and ventilator weaning according to attending physicians
  4. Pain scores and SBS score is noted every 6 hours for the first 24 hours, and every day for the next 24 hours until extubation.
  5. Attending physicians assessed that subject could be weaned: pain scores, SBS score, WAT-1 score
  6. Extubation. Researcher did not take part in the judgement of extubation.

INTERVENTIONS:
Other: Sedation and ventilator weaning protocol — Subjects randomized to this group will underwent sedation and ventilator weaning protocol as mentioned before.
  Arms: Sedation and Ventilator Weaning Protocol

SUMMARY:
This research is a single-blinded, randomized controlled trial involving mechanically ventilated children in Pediatric Intensive Care Unit, Cipto Mangunkusumo Hospital, Indonesia. Subjects were divided into two groups: intervention vs control group. Primary and secondary outcomes will be measure pre, during, and post treatment.

DETAILED DESCRIPTION:
As of today, there is no sedation and ventilator weaning protocol in our PICU. Decision for sedation and ventilator weaning were based on attending physicians clinical judgement, which greatly varies among individual. Previous study on the use of these protocols showed a favorable outcome. We aim to assess the safety and effectiveness of this protocol in our PICU.

Subjects were recruited consecutively and randomized into intervention and control group.

* Intervention group: sedation and ventilator weaning protocol
* Control group: no protocol

Primary outcomes:

* FLACC score
* COMFORT score
* Ventilator days

Secondary outcomes:

* Self extubation
* Reintubation
* PICU Length of stay
* Frequency of asynchrony
* NIRS value
* VIS score

ELIGIBILITY:
Inclusion Criteria:

* Patient who need mechanical ventilation for more than 12 hours

Exclusion Criteria:

* PICU admission due to post cardiac and respiratory arrest

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Face, Leg, Activity, Cry, Consolability (FLACC) score hour 0 | every 6 hours for the first 24 hours, once daily until extubation. This is the baseline. Once the patient was intubated, FLACC scoring of hour 0 will be assessed and noted.
  Pain scoring. Each characteristic has 0-2 points with maximum 10 points. The greater number indicate greater pain score.
Face, Leg, Activity, Cry, Consolability (FLACC) score hour 6 | FLACC scoring of hour 6 will be measured 6 hours after hour 0 was measured. Hour 6 is measured from the time the subject was intubated.
  Pain scoring. Each characteristic has 0-2 points with maximum 10 points. The greater number indicate greater pain score.
Face, Leg, Activity, Cry, Consolability (FLACC) score hour 12 | FLACC scoring of hour 12 will be measured 12 hours after hour 0 was measured. Hour 12 is measured from the time the subject was intubated.
  Pain scoring. Each characteristic has 0-2 points with maximum 10 points. The greater number indicate greater pain score.
Face, Leg, Activity, Cry, Consolability (FLACC) score hour 18 | FLACC scoring of hour 18 will be measured 18 hours after hour 0 was measured. Hour 18 is measured from the time the subject was intubated.
  Pain scoring. Each characteristic has 0-2 points with maximum 10 points. The greater number indicate greater pain score.
Face, Leg, Activity, Cry, Consolability (FLACC) score day 1 until extubation | Scoring will be assessed every morning. If the subject was intubated at night, scoring for day 1 will be measured in the morning the day after tomorrow. Thereafter, the measurement will be taken every morning, 24 hour apart until the subject extubation.
  Pain scoring. Each characteristic has 0-2 points with maximum 10 points. The greater number indicate greater pain score.
Face, Leg, Activity, Cry, Consolability (FLACC) score extubation day | This score will be taken when the subject was stopped from all sedative and analgetics, just before extubation. Monitoring of extubation will be conducted until 56 days after initial intubation.
  Pain scoring. Each characteristic has 0-2 points with maximum 10 points. The greater number indicate greater pain score.
COMFORT score hour 0 | This is the baseline. Once the patient was intubated, COMFORT scoring of hour 0 will be assessed and noted.
  Sedation scoring. It consists of 8 components. Each component has a score of 1-5, max score 40. Scores of 8 - 17 are over-sedated, scores between 17 - 26 are adequately sedated, and scores between 27 - 40 are under-sedated
COMFORT score hour 6 | COMFORT scoring of hour 6 will be measured 6 hours after hour 0 was measured. Hour 6 is measured from the time the subject was intubated.
  Sedation scoring. It consists of 8 components. Each component has a score of 1-5, max score 40. Scores of 8 - 17 are over-sedated, scores between 17 - 26 are adequately sedated, and scores between 27 - 40 are under-sedated
COMFORT score hour 12 | COMFORT scoring of hour 12 will be measured 12 hours after hour 0 was measured. Hour 12 is measured from the time the subject was intubated.
  Sedation scoring. It consists of 8 components. Each component has a score of 1-5, max score 40. Scores of 8 - 17 are over-sedated, scores between 17 - 26 are adequately sedated, and scores between 27 - 40 are under-sedated
COMFORT score hour 18 | COMFORT scoring of hour 18 will be measured 18 hours after hour 0 was measured. Hour 18 is measured from the time the subject was intubated.
  Sedation scoring. It consists of 8 components. Each component has a score of 1-5, max score 40. Scores of 8 - 17 are over-sedated, scores between 17 - 26 are adequately sedated, and scores between 27 - 40 are under-sedated
COMFORT score day 1 until extubation | Scoring will be assessed every morning. If the subject was intubated at night, scoring for day 1 will be measured in the morning the day after tomorrow. Thereafter, the measurement will be taken every morning, 24 hour apart until the subject extubation.
  Sedation scoring. It consists of 8 components. Each component has a score of 1-5, max score 40. Scores of 8 - 17 are over-sedated, scores between 17 - 26 are adequately sedated, and scores between 27 - 40 are under-sedated
COMFORT score extubation day | This score will be taken when the subject was stopped from all sedative and analgetics, just before extubation. Monitoring of extubation will be conducted until 56 days after initial intubation.
  Sedation scoring. It consists of 8 components. Each component has a score of 1-5, max score 40. Scores of 8 - 17 are over-sedated, scores between 17 - 26 are adequately sedated, and scores between 27 - 40 are under-sedated
Ventilator time | From intubation to extubation which would not need reintubation within 48 hours of extubation, measurement of the time frame may be assessed up to 28 days measured from intubation time.
  Time to extubation (days)

SECONDARY OUTCOMES:
Reintubation frequency | Frequency of subject who are extubated to be reintubated within 48 hours after extubation. Assessment will be noted up to 28 days measured from the first time intubation was performed.
  Number of times subject was reintubated within 48 hours after extubation
Self extubation frequency | Frequency of self extubation by the patient during one episode of intubation. Assessment will be noted up to 28 days measured from the first time intubation was performed.
  Number of times subject was self extubated during one episode of intubation
PICU length of stay | Length of stay in PICU from admission until patient's death or step-down to the pediatric ward. Assessment of PICU length of stay will be noted up to 56 days measured from the first day of PICU admission as day 1.
  Days from PICU admission to death or move outside the PICU to the ward
Near infrared spectroscopy minute 5 | The scoring will be noted during minute-5 after sedatives/analgetic administration following intubation.
  Value of Near infrared spectroscopy (NIRS) during minute 5 after administration of sedatives or analgetic. NIRS values of less than 40% for 10 minutes or a 20% decrease from baseline indicated anaerobic metabolism and ischemic brain injury.
Near infrared spectroscopy hour-1 | The scoring will be noted during hour-1 after sedatives/analgetic administration following intubation.
  Value of Near infrared spectroscopy (NIRS) during minute 5 after administration of sedatives or analgetic. NIRS values of less than 40% for 10 minutes or a 20% decrease from baseline indicated anaerobic metabolism and ischemic brain injury.
Near infrared spectroscopy hour-6 | The scoring will be noted during hour-6 after sedatives/analgetic administration following intubation.
  Value of Near infrared spectroscopy (NIRS) during minute 5 after administration of sedatives or analgetic. NIRS values of less than 40% for 10 minutes or a 20% decrease from baseline indicated anaerobic metabolism and ischemic brain injury.
Near infrared spectroscopy hour-12 | The scoring will be noted during hour-12 after sedatives/analgetic administration following intubation.
  Value of Near infrared spectroscopy (NIRS) during minute 5 after administration of sedatives or analgetic. NIRS values of less than 40% for 10 minutes or a 20% decrease from baseline indicated anaerobic metabolism and ischemic brain injury.
Inotropic intervention | The inotropic intervention will be noted throughout PICU admission up to 14 days of mechanical ventilation days.
  All inotropes used will be noted as secondary outcome to identify the hypotensive and/or bradycardia complications that might be caused due to usage of sedatives and analgesia. The usage will be divided into two categories: Yes and No usage of inotrope
Vasoactive-Inotropic Score | The VIS score will be measured once during PICU admission up to 14 days of mechanical ventilation days.. The highest value will be recorded and categorized into two groups
  The VIS were extracted from the formula: dopamine dose (μg/kg/minute) + dobutamine dose (μg/kg/minute) + 100 x epinephine dose (μg/kg/minute) + 10 x milrinone dose (μg/kg/minute) + 10,000 x vasopressine dose (unit/kg/minute) + 100 x norepinefrine dose (μg/kg/minute). The VIS score was categorized into two (≥20 dan <20).

CONTACTS AND LOCATIONS:
Overall Officials: Antonius H. Pudjiadi, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No